CLINICAL TRIAL: NCT02533063
Title: Semi-Recumbent Vibration Therapy in Older Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 2015-0480
Record Dates: First submitted 2015-08-19; First posted 2015-08-26 (Estimated); Results first posted 2019-04-02 (Actual); Last update posted 2019-04-02 (Actual); Status verified 2019-03

CONDITIONS: Sarcopenia; Aging
MeSH Terms: conditions — Sarcopenia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Combination Treatment (Active Comparator): In the "loading + vibration group" (intervention group), subjects will be seated in the VibeTech One system and vibratory acceleration will be 30Hz and the applied load will be 50% of body weight up to a device maximum applied load of 100 lbs. Vibration intensity will initially be set to 0.2 g and will increase by 0.2 g every other week, as tolerated by the subject, and max out at 1.0 g.
  Interventions: Device: VibeTech One
- Sham Treatment (Sham Comparator): In the "loading only" group (control group) participants will be seated in the vibration device (VibeTech One) and will experience loading of their leg muscles through the device.
  Interventions: Device: VibeTech One

INTERVENTIONS:
Device: VibeTech One — Vibration Training The VibeTech One Rehab Chair allows vibration exercise while seated. A force is applied on a footplate that simulates the weight of standing or partial bodyweight. The participants will train for 10 minutes 3 days per week. In the "loading + vibration group" (intervention group) vibratory acceleration will be 30Hz and the applied load will be 50% of body weight up to a device maximum applied load of 100 lbs. Vibration intensity will initially be set to 0.2 g and will increase by 0.2 g every other week, as tolerated by the subject, and max out at 1.0 g.

SUMMARY:
This proposed prospective study will evaluate whether a novel exercise approach, seated vibration therapy, can improve function in the target population of older adults. Therefore, the primary aim of this pilot is to examine the effect of vibration therapy on muscle function (balance, muscle power and strength) and muscle mass.

DETAILED DESCRIPTION:
There are four study visits; screening/baseline followed by eight weeks of training three times a week, visit 1 at eight weeks followed by 4 weeks of washout, Visit 2 at 12 weeks followed by eight weeks of training three times a week, and a final Visit 3 at 20 weeks.

At the screening visit, volunteers will be asked to perform tests included in the short physical performance battery (SPPB) (gait speed, chair rise, balance). If the participants score is ≤ 9 or ≤ 2 in any of the three tests included in the SPPB they will be eligible for the intervention phase. At the baseline visit several questionnaires will be obtained and participants then will proceed with muscle function tests (SPPB, jumping mechanography, grip strength, timed-up-and-go test).

Participants will then be randomized into one of two groups. The first group will receive vibration + loading treatment for the first 8 weeks, the second group will receive sham treatment (loading only). After 8 weeks both groups will go through a 4 week wash-out period and then crossover will occur. The first group will now receive sham treatment (loading only) while the second group will receive vibration + loading treatment. The participants will train for 10 minutes, 3 times a week, during the active 16 total weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women age ≥ 70 years
2. Able and willing to sign informed consent
3. Able to stand without assistance
4. Able and willing to train for 10 minutes, 3 times per week
5. Total SPPB score of ≤ 9 or ≤ 2 in any of the three tests included in the SPPB

Exclusion Criteria:

1. Cognitive impairment to the degree that it limits the ability of signing informed consent
2. Unable to sit upright for 10 minutes
3. History of injury or surgery within the prior six months which limits the ability to ambulate
4. Major illness that might cause missed training sessions or visits.

Min Age: 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 32 (Actual)
Dates: Start 2015-11; Primary Completion 2017-02-15 (Actual); Study Completion 2017-02-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bjoern Buehring, M.D., Principal Investigator — University of Wisconsin, Madison
Locations (1):
- Jewish Home and Care Center, Milwaukee, Wisconsin, United States

REFERENCES:
- [Derived] Taani MH, Binkley N, Gangnon R, Krueger D, Buehring B. Effect of semi-recumbent vibration exercise on muscle outcomes in older adults: a pilot randomized controlled clinical trial. BMC Geriatr. 2022 Apr 18;22(1):335. doi: 10.1186/s12877-022-03052-0. PMID 35436920

RESULTS

PARTICIPANT FLOW:
Groups:
- Loading + Vibration, Then Loading Only; Loading Only, Then Loading + Vibration: In "Loading + Vibration" phase, subjects will be seated in the VibeTech One Rehab Chair, which allows vibration exercise while seated. A force is applied on a footplate that simulates the weight of standing or partial bodyweight. The participants will train for 10 minutes 3 days per week. The vibratory acceleration will be 30Hz and the applied load will be 50% of body weight up to a device maximum applied load of 100 lbs. Vibration intensity will initially be set to 0.2 g and will increase by 0.2 g every other week, as tolerated by the subject, and max of 1.0 g.
  In "Loading Only" phase participants will be seated in the vibration device (VibeTech One) and will experience loading of their leg muscles through the device with no vibration.
  There will be a four week washout period between the two interventions.
Period: Intervention 1 (8 Weeks)
Arm/Group | Loading + Vibration, Then Loading Only | Loading Only, Then Loading + Vibration
Started | 16 | 16
Completed | 14 | 11
Not Completed | 2 | 5
Period: Washout (4 Weeks)
Arm/Group | Loading + Vibration, Then Loading Only | Loading Only, Then Loading + Vibration
Started | 14 | 11
Completed | 14 | 11
Not Completed | 0 | 0
Period: Intervention 2 (8 Weeks)
Arm/Group | Loading + Vibration, Then Loading Only | Loading Only, Then Loading + Vibration
Started | 14 | 11
Completed | 14 | 11
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Loading + Vibration, Then Loading Only; Loading Only, Then Loading + Vibration: In "Loading + Vibration" intervention phase, subjects will be seated in the VibeTech One Rehab Chair, which allows vibration exercise while seated. A force is applied on a footplate that simulates the weight of standing or partial bodyweight. The participants will train for 10 minutes 3 days per week. The vibratory acceleration will be 30Hz and the applied load will be 50% of body weight up to a device maximum applied load of 100 lbs. Vibration intensity will initially be set to 0.2 g and will increase by 0.2 g every other week, as tolerated by the subject, and max of 1.0 g.
  In "Loading Only" control phase participants will be seated in the vibration device (VibeTech One) and will experience loading of their leg muscles through the device with no vibration.
- Total: Total of all reporting groups
Arm/Group | Loading + Vibration, Then Loading Only | Loading Only, Then Loading + Vibration | Total
Number analyzed (Participants) | 16 | 16 | 32
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 16 | 16 | 32
Age, Continuous [Mean (Full Range); unit: years] | 87.9 [74.9 to 99.0] | 86.9 [75.7 to 86.9] | 87.4 [74.9 to 99.0]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 13 | 23
  Male | 6 | 3 | 9
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 16 | 16 | 32
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 16 | 16 | 32

OUTCOME MEASURES:

1. Primary Outcome: Weight Corrected Jump Power Based on Participant's Jump on the Jump Force Plate
Description: The primary aim of this pilot is to examine the effect of vibration therapy on muscle function. Weight corrected jump power will be the main outcome variable. Countermovement jumps are performed on a Leonardo force plate (Novotec Medical, Pforzheim, Germany) following standard procedures. Jumping mechanography uses maximal countermovement jumps to quantitatively measure muscle strength in the legs. Participants will be asked to perform three countermovement jumps. Participants are asked to try to jump as high as possible using both legs. Three jumps are performed; the jump with the highest jump height is used for analysis.
Time Frame: This was collected 4 times: Baseline, after 8 week loading/loading+ vibration training, after 4 week washout, after 8 week crossover training.
Population: In this frail population a number of individuals were unable to perform satisfactory jumps to collect valid data with the current software.
Measure: Mean (Standard Deviation); unit: W/kg
Groups:
- Loading + Vibration: In "Loading + Vibration" intervention phase, subjects will be seated in the VibeTech One Rehab Chair, which allows vibration exercise while seated. A force is applied on a footplate that simulates the weight of standing or partial bodyweight. The participants will train for 10 minutes 3 days per week. The vibratory acceleration will be 30Hz and the applied load will be 50% of body weight up to a device maximum applied load of 100 lbs. Vibration intensity will initially be set to 0.2 g and will increase by 0.2 g every other week, as tolerated by the subject, and max of 1.0 g.
  There will be a four week washout period between the two interventions.
- Loading Only: In "Loading Only" control phase participants will be seated in the vibration device (VibeTech One) and will experience loading of their leg muscles through the device with no vibration. A force is applied on a footplate that simulates the weight of standing or partial bodyweight. The participants will train for 10 minutes 3 days per week.
  There will be a four week washout period between the two interventions.
Arm/Group | Loading + Vibration | Loading Only
Number analyzed (Participants) | 13 | 13
W/kg
  Pre Intervention | 10.53 (5.66) | 10.28 (7.11)
  Post Intervention | 11.10 (7.03) | 8.98 (5.33)
Statistical Analysis 1: Comparison: Loading + Vibration vs Loading Only; Test type: Superiority; p = 0.217, ANOVA

2. Secondary Outcome: Grip Strength
Description: Grip Strengthwas acquired using a JAMAR hand dynamometer in the routine clinical manner. Measurements were recorded using participants' non-dominant hand and repeated 3 times to determine maximum grip strength.
Time Frame: Measured at Baseline, after Intervention 1, after Washout, and after Intervention 2.
Measure: Mean (Standard Deviation); unit: Force (kg)
Arm/Group | Loading + Vibration | Loading Only
Number analyzed (Participants) | 25 | 25
Force (kg)
  Pre Intervention | 13.8 (6.0) | 12.9 (5.6)
  Post Intervention | 13.3 (6.4) | 14.1 (5.0)
Statistical Analysis 1: Comparison: Loading + Vibration vs Loading Only; Test type: Superiority; p = 0.501, ANOVA

3. Secondary Outcome: Gait Speed
Description: Gait speed will be measured by instructing participants to walk four meters at their normal pace; they are timed with a stopwatch. This test will be repeated twice. The walk performed in the least time will be utilized for scoring purposes.
Time Frame: Measured at Baseline, after Intervention 1, after Washout, and after Intervention 2.
Measure: Mean (Standard Deviation); unit: Speed (m/sec)
Groups:
- Loading + Vibration: In "Loading + Vibration" intervention phase, subjects will be seated in the VibeTech One Rehab Chair, which allows vibration exercise while seated. A force is applied on a footplate that simulates the weight of standing or partial bodyweight. The participants will train for 10 minutes 3 days per week. The vibratory acceleration will be 30Hz and the applied load will be 50% of body weight up to a device maximum applied load of 100 lbs. Vibration intensity will initially be set to 0.2 g and will increase by 0.2 g every other week, as tolerated by the subject, and max of 1.0 g.
  In "Loading Only" control phase participants will be seated in the vibration device (VibeTech One) and will experience loading of their leg muscles through the device with no vibration.
  There will be a four week washout period between the two interventions.
Arm/Group | Loading + Vibration | Loading Only
Number analyzed (Participants) | 25 | 25
Speed (m/sec)
  Pre Intervention | 0.6 (0.2) | 0.7 (0.2)
  Post Intervention | 0.7 (0.3) | 0.7 (0.2)
Statistical Analysis 1: Comparison: Loading + Vibration vs Loading Only; Test type: Superiority; p = 0.151, ANOVA

4. Secondary Outcome: Sway
Description: Sway is assessed by having the participants stand with feet being placed side by side for ten seconds. Participants will be wearing MobilityLabTM (APDM, Portland, OR) sensors on their chest, lower back, wrists and feet during these tests to collect computerized sway data.
Time Frame: Measured at Baseline, after Intervention 1, after Washout, and after Intervention 2.
Population: Not all participants could complete the balance exercise and provide valid data for this measure.
Measure: Mean (Standard Deviation); unit: Area (cm square)
Arm/Group | Loading + Vibration | Loading Only
Number analyzed (Participants) | 10 | 10
Area (cm square)
  Pre Intervention | 9.2 (15.8) | 4.8 (6.3)
  Post Intervention | 5.8 (3.4) | 4.7 (4.2)
Statistical Analysis 1: Comparison: Loading + Vibration vs Loading Only; Test type: Superiority; p = 0.450, ANOVA

5. Secondary Outcome: Short Physical Performance Battery (SPPB)
Description: The short physical performance battery (SPPB) consists of gait speed as determined by a four-meter walk, timed repeated chair rise and standing balance. Gait speed will be measured by instructing participants to walk four meters at their normal pace; timed with a stopwatch and is repeated twice. The walk performed in the least time will be utilized for SPPB scoring purposes. The timed repeated chair rise has participants stand up from a chair five times without the use of their arms, if possible. Time to complete five stands is measured. Standing balance is assessed by having the participants stand in three positions of increasing difficulty for 10 seconds each. Standardized instructions will be given to all participants and the test performed twice. The SPPB will be conducted and scored in standard manner, score 0-12, with lower scores indicating mobility limitations. Participants will be wearing MobilityLabTM sensors to collect computerized data for these tests.
Time Frame: Measured at Baseline, after Intervention 1, after Washout, and after Intervention 2.
Population: Not all participants completed the SPPB test.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Loading + Vibration | Loading Only
Number analyzed (Participants) | 21 | 21
score on a scale
  Pre Intervention | 6.8 (2.8) | 7.0 (2.8)
  Post Intervention | 6.8 (2.8) | 7.0 (3.0)
Statistical Analysis 1: Comparison: Loading + Vibration vs Loading Only; Test type: Superiority; p = 0.678, ANOVA

6. Secondary Outcome: Timed-Up-and-Go (TUG)
Description: The Timed-Up-and-Go (TUG) test will be performed twice; participants will be seated in an armless chair, upon instruction, they will be asked to stand, which starts the timing, they will walk 3 meters past a mark on the floor at their normal pace, turn around and return to a full seated position, at which time the test will end.
Time Frame: Measured at Baseline, after Intervention 1, after Washout, and after Intervention 2.
Population: Not all participants completed the TUG testing.
Measure: Mean (Standard Deviation); unit: Time (seconds)
Arm/Group | Loading + Vibration | Loading Only
Number analyzed (Participants) | 20 | 20
Time (seconds)
  Pre Intervention | 18.6 (7.8) | 18.4 (6.8)
  Post Intervention | 20.5 (10.1) | 19.3 (8.4)
Statistical Analysis 1: Comparison: Loading + Vibration vs Loading Only; Test type: Superiority; p = 0.060, ANOVA

7. Other Pre Specified Outcome: Adherence and Factors That Influence Adherence-Exercise Enjoyment
Description: Exercise enjoyment for each intervention was assessed using the validated questionnaire, "5-point Likert scale." Response options include "strongly agree", "agree", "neutral", "disagree", "strongly agree".
Time Frame: This was collected at the end of each 8 week intervention period.
Measure: Number; unit: percentage of participants
Arm/Group | Loading + Vibration | Loading Only
Number analyzed (Participants) | 25 | 25
percentage of participants
  Strongly agree | 12 | 0
  Agree to Neutral | 40 | 33
  Neutral | 48 | 67
  Disagree | 0 | 0
  Strongly disagree | 0 | 0

8. Other Pre Specified Outcome: Adherence and Factors That Influence Adherence-Pain
Description: Self-reported pre- and post-training pain during the vibration intervention and control sessions were calculated as the mean for each participant using a validated questionnaire, "Comprehensive Pain Assessment Form" with scale from 0-10, 0 being no pain and 10 being severe pain.
Time Frame: This was collected before and after training during each of the 8 week interventions.
Measure: Number; unit: percentage of participants
Arm/Group | Loading + Vibration | Loading Only
Number analyzed (Participants) | 25 | 25
percentage of participants
  Pre-training 0-3 | 84 | 96
  Pre-training 4-6 | 16 | 4
  Pre-training 7-10 | 0 | 0
  Post-training 0-3 | 88 | 96
  Post-training 4-6 | 12 | 4
  Post-training 7-10 | 0 | 0

9. Secondary Outcome: Bioelectrical Impedance Spectroscopy (BIS)
Description: An ImpediMed SFB7 device (Eight Mile Plains, Queensland, Australia) will be used to obtain these measurements. Participants will be positioned supine for a minimum of 10 minutes prior to acquisition; adequate separation of their legs will be obtained to allow for accurate BIS measurement. Measurements will be obtained by placing four EKG-like electrodes on the skin of the participant's hand, feet and knee. Wires will be attached from the BIS device to these skin electrodes. Painless electric waves will be sent through the tissues as noted above. Each measurement lasts only a few seconds. This method will generate measurements of lean mass.
Time Frame: Measured at Baseline, after Intervention 1, after Washout, and after Intervention 2.
Measure: Mean (Standard Deviation); unit: Mass (kg)
Arm/Group | Loading + Vibration | Loading Only
Number analyzed (Participants) | 21 | 23
Mass (kg)
  Pre Intervention | 41.75 (7.36) | 41.86 (6.34)
  Post Intervention | 42.19 (8.23) | 41.71 (6.71)
Statistical Analysis 1: Comparison: Loading + Vibration vs Loading Only; Test type: Superiority; p = 0.483, ANOVA

ADVERSE EVENTS:
Time Frame: 20 weeks
Groups:
- Loading Only: In "Loading Only" ocntrol phase participants will be seated in the vibration device (VibeTech One) and will experience loading of their leg muscles through the device with no vibration. A force is applied on a footplate that simulates the weight of standing or partial bodyweight. The participants will train for 10 minutes 3 days per week.
  There will be a four week washout period between the two interventions.
Arm/Group | Loading + Vibration | Loading Only
All-Cause Mortality (participants affected / at risk) | 0/32 | 0/32
Serious Adverse Events (participants affected / at risk) | 4/32 | 2/32
Other Adverse Events (participants affected / at risk) | 14/32 | 3/32
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Loading + Vibration (N=32) | Loading Only (N=32)
Stomach pain (Gastrointestinal disorders) | 1 (1) | 0/16 (0)
Reaction to antibiotic (General disorders) | 1 (1) | 0 (0)
Heart attack (Cardiac disorders) | 1 (1) | 1 (1)
GI Bleeding (Gastrointestinal disorders) | 1 (2) | 0 (0) — GI bleeding reported, noted worsening of existing Crohn's disease
Hip fracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Loading + Vibration (N=32) | Loading Only (N=32)
Leg pain (Musculoskeletal and connective tissue disorders) | 12 (12) | 3 (3)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Parkinsons disease (Nervous system disorders) | 0 (0) | 1 (1) — Reported worsening of existing Parkinson's disease sympotoms
Vertebral fracture (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) — Reported fall with thorasic vertebral fracture
Blood clot (Blood and lymphatic system disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-06-01): https://cdn.clinicaltrials.gov/large-docs/63/NCT02533063/Prot_SAP_000.pdf